CLINICAL TRIAL: NCT03834064
Title: Oral Health Promotion Strategy for Persons With Intellectual/Developmental Disabilities
Acronym: OHPROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Himabindu Dukka, Assistant Professor, University of Louisville
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16020E; U01DE025833 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-02-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Oral Health

STUDY DESIGN:
Intervention Model Description: The primary objective of this study is to assess the direct effect of the OHPROM strategy on oral health status of persons with IDD at post intervention [4-month] and sustained [12-month] in comparison to the control group
Who Masked: Outcomes Assessor
Masking Description: The dentist assessing the oral health status of the intervention and control participants will be masked to participant group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Homes where participants with intellectual/developmental disabilities reside will be randomly assigned to the intervention arm. Caregivers working in that home will receive the oral health promotion strategy/intervention over the course of a year.
  Interventions: Behavioral: Oral health promotion strategy
- Control (No Intervention): Homes where participants with intellectual/developmental disabilities reside will be randomly assigned to the control arm. Caregivers in that home will not receive the oral health promotion strategy/intervention over the course of a year but will be offered a compressed intervention after a year.

INTERVENTIONS:
Behavioral: Oral health promotion strategy — The proposed intervention is comprised of four components : (a) planned action including a behavioral contract Activity 1) with caregivers and action planning for oral health (Activity 2), (b) caregiver capacity building with didactic training (Activity 3), observational learning and caregiver practice (Activity 4); (c) environmental adaptations with location of oral health activities and reminder posters - physical environment (Activity 5) and administrative oral health support- (social environment (Activity 6); and (d) reinforcement with caregiver coaching (Activity 7).
  Arms: Intervention

SUMMARY:
A Phase II cluster randomized controlled trial of the (OHPROM) strategy/intervention will be conducted in partnership with several organizations that provide residential services for persons with intellectual developmental disabilities (IDD) in north central Kentucky and southern Indiana. The investigators have identified a purposive sample of group homes, caregivers, and persons with IDD and have the support of these organizations.

DETAILED DESCRIPTION:
The proposed intervention is comprised of four components : (a) planned action including a behavioral contract Activity 1) with caregivers and action planning for oral health (Activity 2), (b) caregiver capacity building with didactic training (Activity 3), observational learning and caregiver practice (Activity 4); (c) environmental adaptations with location of oral health activities and reminder posters - physical environment (Activity 5) and administrative oral health support- (social environment (Activity 6); and (d) reinforcement with caregiver coaching (Activity 7).

ELIGIBILITY:
Inclusion Criteria:

* Persons with IDD: To be eligible to participate in this study, an individual must meet all of the following criteria:

  * Be a resident in a group or family home associated with one of the six partner organizations participating in this study
  * Provide signed and dated informed consent form, to be signed by self or a legally authorized representative (LAR), if one has been appointed
  * Be willing and able to comply with all study procedures and expect to be available for the duration of the study
  * Be aged 18 to 75
  * Have at least six teeth
  * Have diagnosis of mild, moderate, severe, or profound intellectual and/or developmental disability

Caregiver staff: To be eligible to participate in this study, caregiver staff must meet all of the following criteria:

* Work as a direct care staff member in a group/family home
* Provide signed and dated informed consent form
* Be willing to comply with all study procedures and be available for the duration of the study
* Be aged 18 to 75

Exclusion Criteria:

* Persons with IDD: Will be excluded (screen failure) if they are unable to cooperate or refuse the oral examination.
* Caregivers: There are no exclusions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is the change in the oral health status of persons with IDD at 4 months and 12 months in comparison to the control group, after controlling for oral health status at baseline as measured by the Modified Gingival Index. | 12 months
  Primary Outcome Measure the Modified Gingival Index (MGI). The MGI assesses the gingival condition, with scores ranging from 0 (no inflammation) to 4 (severe inflammation). Score range 0-128, higher is worse.
The primary outcome of this study is change in the oral health status of persons with IDD at 4 months and 12 months in comparison to the control group, after controlling for oral health status at baseline as measured by the Community Periodontal Index. | 12 months
  Primary Outcome Measure the Community Periodontal Index (CPI). The CPI assesses periodontal disease from a score of 0 (healthy - absence of periodontal disease) to 4 (deep pockets - severe periodontal disease). Score range 1-40, higher is worse outcome.

SECONDARY OUTCOMES:
Change in caregiver self-efficacy from baseline to 4 months and 12 months in the experimental group compared to the control group of caregivers. | 12 months
  Caregivers will self-report self-efficacy using an adapted version of the 10-item General Self- Efficacy Scale (Schwarzer, 1995). The adaptation was made to the lead-in statement in order to ask about general self-efficacy of Caregivers as they provide support to residents' oral hygiene and dietary practices. Response choices are: Never, Almost, Sometimes, Fairly Often, and Very Often. Score range 0-40, higher is good.
Change in caregiver outcome expectancies from baseline to 4 months and 12 months in the experimental group compared to the control group of caregivers. | 12 months
  Caregivers will self-report outcome expectancies using an adapted version of Kakudate et al.'s (2010) 6-item Outcome Expectancies Scale. Response choices are: Strongly Disagree, Disagree, Agree, and Strongly Agree. Score range 0-48, higher good
Change in caregiver behavioral capability from baseline to 4 months and 12 months in the experimental group compared to the control group of caregivers. | 12 months
  Caregivers will self-report behavioral capability using an adapted version of Pradhan's (2016) Carer Activation Measure. Subscales of confidence (6 items) and skills (5 items) to measure behavioral capability. Response choices are: Strongly Disagree, Disagree, Agree, and Strongly Agree. Score range 0-44, higher is good.
Secondary outcomes are change in caregiver perceptions of environmental influences from baseline to 4 months and 12 months in the experimental group compared to the control group of caregivers. | 12 months
  Caregivers will self-report environmental influences using a caregiver questionnaire developed specifically for this study, which assesses caregiver perceptions of the level of influence physical environmental influences (e.g., placement of posters as daily reminders) and social environmental influences (e.g., administrative support through policies and procedures). This is an 8-item scale. Response choices are: Strongly Disagree, Disagree, Agree, and Strongly Agree. Score range 0-32, higher is good.
Change in Oral hygiene practices of persons with IDD will be measured by a dental oral examination guided by the Simplified Oral Hygiene Index (OHI-S) from baseline to 4 months and 12 months in the experimental group compared to the control group. | 12 months
  The OHI-S has two components: the Debris Index and the Calculus Index. Each of these indices represents numerical determinations ranging from 0 (None) to 3 (Covering 2/3rd of tooth surface) of the amount of debris or calculus found on the preselected tooth surfaces. The six surfaces examined for the OHI-S are selected from four posterior and two anterior teeth. The buccal surfaces of the selected upper molars and the lingual surfaces of the selected lower molars are inspected. In the anterior portion of the mouth, the labial surfaces of the upper right (11) and the lower left central incisors The average individual or group debris and calculus scores are combined to obtain the Simplified Oral Hygiene Index. The CI-S and DI-S values may range from 0 to 3; the OHI-S values from 0 to 6. Higher scores indicate a worse outcome.
Change in oral hygiene practices of persons with IDD will be measured by a caregiver-reported Daily Oral Health Checklist in the experimental group compared to the control group from baseline to 4 months and 12 months. | 12 months
  The Daily Oral Health Checklist will be completed daily by each Caregiver for three days at all three time points in the study. These data will be used to calculate an index to assess Oral Hygiene Practices of residents' use (daily - yes/no) of oral hygiene devices as well as whether adequate time (at least one minute daily) was spent on oral hygiene activities, and whether hygiene activities were completed alone or with caregiver assistance. Dietary practices of persons with IDD will also be measured by the 3-day Daily Oral Health Checklist and completed by Caregivers to assess the frequency and timing of food and beverages that are good and bad for teeth and if caregivers cooperation strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No